CLINICAL TRIAL: NCT01264939
Title: A Phase III, Multicenter, Randomized, Double-blind, Placebo-controlled Safety Study of Xolair (Omalizumab) in Patients With Chronic Idiopathic Urticaria (CIU) Who Remain Symptomatic Despite Treatment With H1 Antihistamines, H2 Blockers, and/or Leukotriene Receptor Antagonists
Brief Title: A Safety Study of Xolair (Omalizumab) in Patients With Chronic Idiopathic Urticaria (CIU) Who Remain Symptomatic Despite Treatment With H1 Antihistamines, H2 Blockers, and/or Leukotriene Receptor Antagonists
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Q4883g; GA00889 (Other: Hoffmann-La Roche)
Record Dates: First submitted 2010-12-20; First posted 2010-12-22 (Estimated); Results first posted 2013-11-26 (Estimated); Last update posted 2013-11-26 (Estimated); Status verified 2013-09

CONDITIONS: Chronic Idiopathic Urticaria
MeSH Terms: conditions — Chronic Urticaria | interventions — Omalizumab; Histamine Antagonists; Leukotriene Antagonists; Diphenhydramine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor

ARMS (2):
- Placebo (Placebo Comparator): Participants received placebo subcutaneously every 4 weeks during the 24 week treatment period.
  Interventions: Drug: Placebo; Drug: H1 antihistamine, H2 antihistamine, leukotriene receptor antagonist; Drug: Diphenhydramine
- Omalizumab 300 mg (Experimental): Participants received omalizumab 300 mg subcutaneously every 4 weeks during the 24 week treatment period.
  Interventions: Drug: Omalizumab; Drug: H1 antihistamine, H2 antihistamine, leukotriene receptor antagonist; Drug: Diphenhydramine

INTERVENTIONS:
Drug: Omalizumab — Omalizumab was supplied as a lyophilized, sterile powder in a single-use vial.
  Other Names: Xolair
  Arms: Omalizumab 300 mg
Drug: Placebo — Placebo was supplied as a lyophilized, sterile powder in a single-use vial without study drug.
  Arms: Placebo
Drug: H1 antihistamine, H2 antihistamine, leukotriene receptor antagonist — Participants were required to maintain stable doses of their pre-randomization combination therapy with an H1 antihistamine and either an H2 blocker or leukotriene receptor antagonist, or all 3 drugs in combination, throughout the 24-week treatment period and 16-week follow-up period of the 40-week study.
Drug: Diphenhydramine — Participants were provided with diphenhydramine 25 mg for itch relief on an as-needed basis, up to a maximum of 3 doses within 24 hours for the duration of the 40-week study.

SUMMARY:
The study is a global Phase III, multicenter, randomized, double-blind, placebo controlled, parallel-group study to evaluate the safety and efficacy of omalizumab administered subcutaneously as an add-on therapy for the treatment of adolescent and adult patients aged 12-75 who have been diagnosed with chronic idiopathic urticaria (CIU) who remain symptomatic despite standard-dosed H1 antihistamine treatment (including doses up to 4 times above the approved dose level), H2 blockers, and/or leukotriene receptor antagonists (LTRA).

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of chronic idiopathic urticaria (CIU) refractory to H1 antihistamines, H2 blockers, and/or leukotriene receptor antagonists (LTRA) at the time of randomization.

  * The presence of itch and hives for > 6 consecutive weeks at any time prior to enrollment despite current use of H1 antihistamine (up to 4 times the approved dosage), H2 blocker, and/or LTRA treatment during this time.
  * Urticaria activity score over 7 days (UAS7) score (range 0-42) ≥ 16 and itch component of UAS7 (range 0-21) ≥ 8 during 7 days prior to randomization (Week 0).
  * In-clinic UAS ≥ 4 on at least one of the screening visit days (Day -14, Day -7, or Day 1).
* For women of childbearing potential, agreement to use an acceptable form of contraception and to continue its use for the duration of the study.

Exclusion Criteria:

* Treatment with an investigational agent within 30 days prior to screening.
* Weight less than 20 kg (44 lbs).
* Clearly defined underlying etiology for chronic urticarias other than CIU.
* Evidence of parasitic infection.
* Atopic dermatitis, bullous pemphigoid, dermatitis herpetiformis, senile pruritus, or other skin disease associated with itch.
* Previous treatment with omalizumab within a year prior to screening.
* Routine doses of the following medications within 30 days prior to screening: Systemic or cutaneous (topical) corticosteroids (prescription or over the counter), hydroxychloroquine, methotrexate, cyclosporine, or cyclophosphamide.
* Intravenous (IV) immunoglobulin G (IVIG), or plasmapheresis within 30 days prior to screening.
* Regular (daily/every other day) doxepin (oral) use within 6 weeks prior to screening.
* Patients with current malignancy, history of malignancy, or currently under work-up for suspected malignancy except non-melanoma skin cancer that has been treated or excised and is considered resolved.
* Hypersensitivity to omalizumab or any component of the formulation.
* History of anaphylactic shock.
* Presence of clinically significant cardiovascular, neurological, psychiatric, metabolic, or other pathological conditions that could interfere with the interpretation of the study results and or compromise the safety of the patients.
* Evidence of current drug or alcohol abuse.

Ages: 12 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 336 (Actual)
Dates: Start 2011-02; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Edward R. Conner, M.D., Study Director — Genentech, Inc.
Locations (68):
- United States (38):
  - Scottsdale, Arizona
  - Mission Viejo, California
  - Napa, California
  - Orange, California
  - Sacramento, California
  - San Diego, California
  - Miami, Florida
  - North Palm Beach, Florida
  - Tampa, Florida
  - Savannah, Georgia
  - Evansville, Indiana
  - Iowa City, Iowa
  - Crescent Springs, Kentucky
  - Owensboro, Kentucky
  - Wheaton, Maryland
  - Brookline, Massachusetts
  - Ann Arbor, Michigan
  - Minneapolis, Minnesota
  - Rochester, Minnesota
  - Bozeman, Montana
  - Missoula, Montana
  - Brick, New Jersey
  - Mineola, New York
  - Rochester, New York
  - High Point, North Carolina
  - Sylvania, Ohio
  - Lake Oswego, Oregon
  - Altoona, Pennsylvania
  - Blue Bell, Pennsylvania
  - Hershey, Pennsylvania
  - Charleston, South Carolina
  - Knoxville, Tennessee
  - Dallas, Texas
  - Katy, Texas
  - San Antonio, Texas
  - Draper, Utah
  - South Burlington, Vermont
  - Richmond, Virginia
- Australia (4):
  - Canberra, Australian Capital Territory
  - Brisbane, Queensland
  - Carlton, Victoria
  - Melbourne, Victoria
- Germany (9):
  - Berlin
  - Cologne
  - Erlangen
  - Freiburg im Breisgau
  - Hamburg
  - Lübeck
  - Mainz
  - Marburg
  - Tübingen
- New Zealand (4):
  - Auckland
  - Beckenham
  - Tauranga
  - Wellington
- Poland (3):
  - Krakow
  - Lodz
  - Warsaw
- Singapore, Singapore
- Switzerland (3):
  - Aarau
  - Bern
  - Sankt Gallen
- United Kingdom (6):
  - Cambridge
  - Leicester
  - London
  - Norwich
  - Oxford
  - Sheffield

REFERENCES:
- [Derived] Ferrer M, Gimenez-Arnau A, Saldana D, Janssens N, Balp MM, Khalil S, Risson V. Predicting Chronic Spontaneous Urticaria Symptom Return After Omalizumab Treatment Discontinuation: Exploratory Analysis. J Allergy Clin Immunol Pract. 2018 Jul-Aug;6(4):1191-1197.e5. doi: 10.1016/j.jaip.2018.04.003. Epub 2018 Apr 12. PMID 29655772
- [Derived] Goldstein S, Gabriel S, Kianifard F, Ortiz B, Skoner DP. Clinical features of adolescents with chronic idiopathic or spontaneous urticaria: Review of omalizumab clinical trials. Ann Allergy Asthma Immunol. 2017 Apr;118(4):500-504. doi: 10.1016/j.anai.2017.02.003. PMID 28390587
- [Derived] Saini SS, Omachi TA, Trzaskoma B, Hulter HN, Rosen K, Sterba PM, Courneya JP, Lackey A, Chen H. Effect of Omalizumab on Blood Basophil Counts in Patients with Chronic Idiopathic/Spontaneous Urticaria. J Invest Dermatol. 2017 Apr;137(4):958-961. doi: 10.1016/j.jid.2016.11.025. Epub 2016 Dec 6. No abstract available. PMID 27939380
- [Derived] Gimenez-Arnau AM, Spector S, Antonova E, Trzaskoma B, Rosen K, Omachi TA, Stull D, Balp MM, Murphy T. Improvement of sleep in patients with chronic idiopathic/spontaneous urticaria treated with omalizumab: results of three randomized, double-blind, placebo-controlled studies. Clin Transl Allergy. 2016 Aug 18;6:32. doi: 10.1186/s13601-016-0120-0. eCollection 2016. PMID 27540466
- [Derived] Zazzali JL, Kaplan A, Maurer M, Raimundo K, Trzaskoma B, Solari PG, Antonova E, Mendelson M, Rosen KE. Angioedema in the omalizumab chronic idiopathic/spontaneous urticaria pivotal studies. Ann Allergy Asthma Immunol. 2016 Oct;117(4):370-377.e1. doi: 10.1016/j.anai.2016.06.024. Epub 2016 Jul 14. PMID 27424128
- [Derived] Casale TB, Bernstein JA, Maurer M, Saini SS, Trzaskoma B, Chen H, Grattan CE, Gimenez-Arnau A, Kaplan AP, Rosen K. Similar Efficacy with Omalizumab in Chronic Idiopathic/Spontaneous Urticaria Despite Different Background Therapy. J Allergy Clin Immunol Pract. 2015 Sep-Oct;3(5):743-50.e1. doi: 10.1016/j.jaip.2015.04.015. Epub 2015 Jun 6. PMID 26054553

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Randomized population: All randomized participants regardless of whether they received any study drug.
  One patient in the placebo group was withdrawn after randomization but before receiving treatment due to an adverse event. This patient is 1 of 18 in this reporting group who did not complete the study.
Period: Overall Study
Arm/Group | Placebo | Omalizumab 300 mg
Started | 84 | 252
Completed | 66 | 224
Not Completed | 18 | 28
Not completed — Adverse Event | 1 | 3
Not completed — Lost to Follow-up | 0 | 3
Not completed — Physician Decision | 1 | 1
Not completed — Patient/Guardian Decision | 8 | 10
Not completed — Disease Progression | 8 | 11

BASELINE CHARACTERISTICS:
Population: Modified intent-to-treat (mITT) population: All randomized participants who received at least 1 dose of study drug. One participant (randomized to placebo) did not receive study drug and was not included in the mITT population.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Omalizumab 300 mg | Total
Number analyzed (Participants) | 83 | 252 | 335
Age Continuous [Mean (Standard Deviation); unit: years] | 44.3 (14.7) | 42.7 (13.9) | 43.1 (14.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 55 | 186 | 241
  Male | 28 | 66 | 94

OUTCOME MEASURES:

1. Secondary Outcome: Change From Baseline to Week 12 in the Weekly Itch Severity Score
Description: The weekly itch severity score is the sum of the daily itch severity scores over 7 days and ranges from 0 to 21. The daily itch severity score is the average of the morning and evening scores on a scale of 0 (none) to 3 (severe). The Baseline weekly itch severity score is the sum of the daily itch severity scores over the 7 days prior to the first treatment. A higher itch severity score indicates more severe itching. A negative change score indicates improvement.
Time Frame: Baseline to Week 12
Population: Modified intent-to-treat population: All randomized patients who received at least 1 dose of study drug.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Placebo | Omalizumab 300 mg
Number analyzed (Participants) | 83 | 252
Units on a scale | -4.01 (5.87) | -8.55 (6.01)
Statistical Analysis 1: Comparison: Placebo vs Omalizumab 300 mg; The null hypothesis was that there was no difference between the placebo and the omalizumab 300 mg groups; Test type: Superiority or Other; p < 0.0001, ANCOVA — Multiplicity plan applied to the efficacy endpoints provided strong control of the type I error rate at 0.05 level by pre-specifying the hierarchical order of the efficacy endpoint tests; Covariates included in the analysis were baseline weekly itch severity score (< 13 vs ≥ 13) and baseline weight (< 80 kg vs ≥ 80 kg); Least squares mean difference = -4.52, 95% CI 2-sided [-5.97 to -3.08]

2. Secondary Outcome: Change From Baseline to Week 12 in the Urticaria Activity Score Over 7 Days (UAS7)
Description: The UAS7 is the sum of the daily urticarial activity scores over 7 days and ranges from 0 to 42. The daily urticarial activity score is the average of the morning and evening urticarial activity scores and ranges from 0 to 6. The urticarial activity score is the sum of ratings on a scale of 0 to 3 (0=none to 3=intense/severe) for (1) the number of wheals (hives) and (2) itch intensity over the previous 12 hours, ranges from 0 to 6, and is measured twice daily (morning and evening). The Baseline score is the sum of the daily urticarial activity scores over the 7 days prior to the first treatment. A higher urticarial activity score indicates more urticaria activity. A negative change score indicates improvement.
Time Frame: Baseline to Week 12
Population: Modified intent-to-treat population: All randomized patients who received at least 1 dose of study drug.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Placebo | Omalizumab 300 mg
Number analyzed (Participants) | 83 | 252
Units on a scale | -8.50 (11.71) | -19.01 (13.15)
Statistical Analysis 1: Comparison: Placebo vs Omalizumab 300 mg; The null hypothesis was that there was no difference between the placebo and the omalizumab 300 mg groups; Test type: Superiority or Other; p < 0.0001, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Covariates included in the analysis were baseline UAS7 (< median vs ≥ median) and baseline weight (< 80 kg vs ≥ 80 kg); Least squares mean difference = -10.02, 95% CI 2-sided [-13.17 to -6.86]

3. Secondary Outcome: Change From Baseline to Week 12 in the Weekly Number of Hives Score
Description: The weekly hives score is the sum of the daily hives scores over 7 days and ranges from 0 to 21. The number of hives is measured twice daily (morning and evening) on a scale of 0 (none) to 3 (> 12 hives per 12 hours). The daily hives score is the average of the morning and evening scores. The Baseline score is the sum of the daily hives scores over the 7 days prior to the first treatment. A higher score indicates more hives. A negative change score indicates improvement.
Time Frame: Baseline to Week 12
Population: Modified intent-to-treat population: All randomized patients who received at least 1 dose of study drug.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Placebo | Omalizumab 300 mg
Number analyzed (Participants) | 83 | 252
Units on a scale | -4.49 (6.33) | -10.46 (7.74)
Statistical Analysis 1: Comparison: Placebo vs Omalizumab 300 mg; The null hypothesis was that there was no difference between the placebo and the omalizumab 300 mg groups; Test type: Superiority or Other; p < 0.0001, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Covariates included in the analysis were baseline weekly number of hives score (< median vs ≥ median) and baseline weight (< 80 kg vs ≥ 80 kg); Least squares mean difference = -5.90, 95% CI 2-sided [-7.72 to -4.07]

4. Secondary Outcome: Time to Minimally Important Difference (MID) Response in the Weekly Itch Severity Score by Week 12
Description: The time to the MID response is the number of weeks from the start of treatment (Baseline) until the time point at which the first MID response occurs. The MID response is defined as a reduction ≥ 5 points from Baseline in the weekly itch severity score. The weekly itch severity score is the sum of the daily itch severity scores over 7 days and ranges from 0 to 21. The daily itch severity score is the average of the morning and evening scores on a scale of 0 (none) to 3 (severe). The Baseline weekly itch severity score is the sum of the daily itch severity scores over the 7 days prior to the first treatment. A higher itch severity score indicates more severe itching.
Time Frame: Baseline to Week 12
Population: Modified intent-to-treat population: All randomized patients who received at least 1 dose of study drug. Only patients with a MID response were included in the analysis.
Measure: Median (95% Confidence Interval); unit: Weeks
Arm/Group | Placebo | Omalizumab 300 mg
Number analyzed (Participants) | 83 | 252
Weeks | 5.0 [3.0 to 7.0] | 2.0 [1.0 to 2.0]
Statistical Analysis 1: Comparison: Placebo vs Omalizumab 300 mg; The null hypothesis was that there was no difference between the placebo and the omalizumab 300 mg groups; Test type: Superiority or Other; p < 0.0001, Cox proportional hazards model — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 1, analysis 1]; Hazard Ratio (HR) = 1.99, 95% CI 2-sided [1.47 to 2.68]

5. Secondary Outcome: Percentage of Participants With a UAS7 Score ≤ 6 at Week 12
Description: The UAS7 is the sum of the daily urticarial activity scores over 7 days and ranges from 0 to 42. The daily urticarial activity score is the average of the morning and evening urticarial activity scores and ranges from 0 to 6. The urticarial activity score is the sum of ratings on a scale of 0 to 3 (0=none to 3=intense/severe) for (1) the number of wheals (hives) and (2) itch intensity over the previous 12 hours, ranges from 0 to 6, and is measured twice daily (morning and evening). The Baseline score is the sum of the daily urticarial activity scores over the 7 days prior to the first treatment. A higher urticarial activity score indicates more urticaria activity.
Time Frame: Week 12
Population: Modified intent-to-treat population: All randomized patients who received at least 1 dose of study drug.
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo | Omalizumab 300 mg
Number analyzed (Participants) | 83 | 252
Percentage of participants | 12.0 | 52.4
Statistical Analysis 1: Comparison: Placebo vs Omalizumab 300 mg; The null hypothesis was that there was no difference between the placebo and the omalizumab 300 mg groups; Test type: Superiority or Other; p < 0.0001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 1]; Covariates included in the analysis were baseline UAS7 (< median vs ≥ median) and baseline weight (< 80 kg vs ≥ 80 kg)

6. Secondary Outcome: Percentage of Weekly Itch Severity Score MID Responders at Week 12
Description: The percentage of participants with an itch severity score at 12 Weeks at least 5 points lower than at Baseline. The weekly itch severity score is the sum of the daily itch severity scores over 7 days and ranges from 0 to 21. The daily itch severity score is the average of the morning and evening scores on a scale of 0 (none) to 3 (severe). The Baseline weekly itch severity score is the sum of the daily itch severity scores over the 7 days prior to the first treatment. A higher itch severity score indicates more severe itching.
Time Frame: Baseline to Week 12
Population: Modified intent-to-treat population: All randomized patients who received at least 1 dose of study drug.
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo | Omalizumab 300 mg
Number analyzed (Participants) | 83 | 252
Percentage of participants | 39.8 | 69.8
Statistical Analysis 1: Comparison: Placebo vs Omalizumab 300 mg; The null hypothesis was that there was no difference between the placebo and the omalizumab 300 mg groups; Test type: Superiority or Other; p < 0.0001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 1, analysis 1]

7. Secondary Outcome: Change From Baseline to Week 12 in the Weekly Size of the Largest Hive Score
Description: The weekly size of the largest hive score is the sum of the daily size of the largest hive scores over 7 days and ranges from 0 to 21. The daily size of the largest hive score is assessed twice daily (morning and evening) on a scale of 0 (none) to 3 (> 2.5 cm). The daily size of the largest hive score is the average of the morning and evening scores. The Baseline weekly size of the largest hive score is calculated over the 7 days prior to the first treatment. A higher score indicates larger hives. A negative change score indicates a reduction in hive size.
Time Frame: Baseline to Week 12
Population: Modified intent-to-treat population: All randomized patients who received at least 1 dose of study drug.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Placebo | Omalizumab 300 mg
Number analyzed (Participants) | 83 | 252
Units on a scale | -3.09 (5.46) | -8.82 (7.23)
Statistical Analysis 1: Comparison: Placebo vs Omalizumab 300 mg; The null hypothesis was that there was no difference between the placebo and the omalizumab 300 mg groups; Test type: Superiority or Other; p < 0.0001, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Covariates included in the analysis were baseline weekly size of largest hive score (< median vs ≥ median) and baseline weight (< 80 kg vs ≥ 80 kg); Least squares mean difference = -5.61, 95% CI 2-sided [-7.25 to -3.96]

8. Secondary Outcome: Change From Baseline in the Overall Dermatology Life Quality Index (DLQI) Score at Week 12
Description: The DLQI is a 10-item dermatology-specific health-related quality of life measure. Patients rated their dermatology symptoms as well as the impact of their skin condition on various aspects of their lives on a scale of 0 (Not at all) to 3 (Very much). The overall DLQI is the sum of the responses to the 10 items and ranges from 0 to 30. A lower score indicates a better quality of life. A negative change score indicates improvement.
Time Frame: Baseline to Week 12
Population: Modified intent-to-treat population: All randomized patients who received at least 1 dose of study drug and who had a DLQI score at Week 12.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Placebo | Omalizumab 300 mg
Number analyzed (Participants) | 64 | 216
Units on a scale | -5.11 (7.53) | -9.69 (6.85)
Statistical Analysis 1: Comparison: Placebo vs Omalizumab 300 mg; The null hypothesis was that there was no difference between the placebo and the omalizumab 300 mg groups; Test type: Superiority or Other; p < 0.0001, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Covariates included in the analysis were baseline overall DLQI score (< median vs ≥ median) and baseline weight (< 80 kg vs ≥ 80 kg); Least squares mean difference = -4.67, 95% CI 2-sided [-6.28 to -3.06]

9. Secondary Outcome: Percentage of Angioedema-free Days From Week 4 to Week 12
Description: The percentage of angioedema-free days from Weeks 4 to 12 was defined as the number of days for which a patient responded "No" to the angioedema question in the daily diary divided by the total number of days with a non-missing diary entry, starting at the Week 4 visit and ending the day prior to the Week 12 visit.
Time Frame: Week 4 to Week 12
Population: Modified intent-to-treat population: All randomized patients who received at least 1 dose of study drug. Patients who withdrew before the Week 4 visit or who had missing responses for more than 40% of the daily diary entries between the Week 4 visit and the Week 12 visit were not included in the analysis.
Measure: Mean (Standard Deviation); unit: Percentage of days
Arm/Group | Placebo | Omalizumab 300 mg
Number analyzed (Participants) | 68 | 224
Percentage of days | 88.1 (18.9) | 91.0 (21.0)
Statistical Analysis 1: Comparison: Placebo vs Omalizumab 300 mg; The null hypothesis was that there was no difference between the placebo and the omalizumab 300 mg groups; Test type: Superiority or Other; p = 0.0006, Stratified Wilcoxon — [p-value comment as in outcome 1, analysis 1]; Stratification variables included in the analysis were presence of angioedema at baseline (yes vs no) and baseline weight (< 80 kg vs ≥ 80 kg)

10. Secondary Outcome: Percentage of Complete Responders (UAS7 = 0) at Week 12
Description: A complete responder was defined as a participant with a UAS7 score = 0 at Week 12. The UAS7 is the sum of the daily urticarial activity scores over 7 days and ranges from 0 to 42. The daily urticarial activity score is the average of the morning and evening urticarial activity scores and ranges from 0 to 6. The urticarial activity score is the sum of ratings on a scale of 0 to 3 (0=none to 3=intense/severe) for (1) the number of wheals (hives) and (2) itch intensity over the previous 12 hours, ranges from 0 to 6, and is measured twice daily (morning and evening). The Baseline score is the sum of the daily urticarial activity scores over the 7 days prior to the first treatment. A higher urticarial activity score indicates more urticaria activity.
Time Frame: Week 12
Population: Modified intent-to-treat population: All randomized patients who received at least 1 dose of study drug.
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo | Omalizumab 300 mg
Number analyzed (Participants) | 83 | 252
Percentage of participants | 4.8 | 33.7
Statistical Analysis 1: Comparison: Placebo vs Omalizumab 300 mg; The null hypothesis was that there was no difference between the placebo and the omalizumab 300 mg groups; Test type: Superiority or Other; p < 0.0001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 1]; Covariates included in the analysis were baseline UAS7 (< median vs ≥ median) and baseline weight (< 80 kg vs ≥ 80 kg)

11. Primary Outcome: Percentage of Participants With Adverse Events
Description: The percentage of participants with serious adverse events and other adverse events is summarized by MedDRA preferred terms and organ classes in the Reported Adverse Events section below.
Time Frame: Baseline to the end of study (up to 40 weeks)
Population: Safety population: All randomized participants who received at least 1 dose of study drug.
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo | Omalizumab 300 mg
Number analyzed (Participants) | 83 | 252
Percentage of participants | 78.3 | 83.7

ADVERSE EVENTS:
Time Frame: Adverse events were reported that started on or after the first treatment date through the end of the study (up to 40 weeks).
Description: Safety population: All randomized participants who received at least 1 dose of study drug.
  Multiple occurrences of a specific adverse event for a patient were counted once in the frequency for the adverse event.
Arm/Group | Placebo | Omalizumab 300 mg
Serious Adverse Events (participants affected / at risk) | 5/83 | 18/252
Other Adverse Events (participants affected / at risk) | 41/83 | 142/252
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=83) | Omalizumab 300 mg (N=252)
Angina unstable (Cardiac disorders) | 1 | 0
Gastric ulcer (Gastrointestinal disorders) | 0 | 1
Gastritis erosive (Gastrointestinal disorders) | 0 | 1
Cholelithiasis (Hepatobiliary disorders) | 0 | 1
Hypersensitivity (Immune system disorders) | 1 | 0
Gastroenteritis (Infections and infestations) | 0 | 1
Retroperitoneal infection (Infections and infestations) | 0 | 1
Gastroenteritis viral (Infections and infestations) | 0 | 1
Viral infection (Infections and infestations) | 0 | 1
Pelvic abscess (Infections and infestations) | 0 | 1
Lower respiratory tract infection (Infections and infestations) | 0 | 1
Urinary tract infection (Infections and infestations) | 0 | 1
Multiple drug overdose (Injury, poisoning and procedural complications) | 0 | 1
Blood glucose increased (Investigations) | 0 | 1
Blood pressure increased (Investigations) | 0 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 | 1
Depression (Psychiatric disorders) | 0 | 1
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Angioedema (Skin and subcutaneous tissue disorders) | 1 | 4
Urticaria (Skin and subcutaneous tissue disorders) | 1 | 2
Idiopathic urticaria (Skin and subcutaneous tissue disorders) | 0 | 1
Intermittent claudication (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=83) | Omalizumab 300 mg (N=252)
Nausea (Gastrointestinal disorders) | 5 | 15
Diarrhoea (Gastrointestinal disorders) | 5 | 13
Sinusitis (Infections and infestations) | 9 | 31
Nasopharyngitis (Infections and infestations) | 8 | 30
Upper respiratory tract infection (Infections and infestations) | 4 | 29
Urinary tract infection (Infections and infestations) | 1 | 15
Headache (Nervous system disorders) | 6 | 27
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 7 | 11
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 5 | 3
Idiopathic urticaria (Skin and subcutaneous tissue disorders) | 10 | 37
Urticaria (Skin and subcutaneous tissue disorders) | 3 | 14

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.